CLINICAL TRIAL: NCT04766593
Title: Effects of a Specific Programme for the Recovery of Autonomy Plus Multimodal Physical Exercise on Functionality, Physical Performance, and Respiratory Parameters in Oncology Patients With Dyspnoea
Brief Title: Effects of a Specific Programme for the Recovery of Autonomy Plus Multimodal Physical Exercise in Oncology Patients With Dyspnoea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eduardo J Fernández Rodríguez, PhD, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI 2020 07 547
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cancer; Dyspnea
Keywords: Cancer; Rehabilitation; Occupational therapy; Dyspnea; Physical exercise
MeSH Terms: conditions — Neoplasms; Dyspnea; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oncological functional reeducation program (Experimental): It will consist of the following actions:
  1. Prescription of multimodal physical exercise: This therapeutic measure will be carried out both in the individuals of the experimental group and in those of the control group. It will be held daily in two short sessions of 15-20 minutes, one in the morning and one in the afternoon. The sessions were structured according to the recommendations of the American College of Sports Medicine (ACSM) 18, with an initial warm-up (2-3 minutes), a main part (8-12 minutes) and a final cool-down and relaxation (5 minutes).
  2. Retraining in activities of daily living: Gradation and simplification of activities and training in energy saving techniques (EAT).
  Finally, an exhaustive daily record of the activity carried out by the patient will be carried out, from which it will be modified, adapting it to the clinical situation of the patient.
  Interventions: Other: Oncological functional reeducation program
- Prescription of multimodal physical exercise (Active Comparator): This therapeutic measure will be carried out both in the individuals of the experimental group and in those of the control group. It will be held daily in two short sessions of 15-20 minutes, one in the morning and one in the afternoon. The guideline will be to maintain a multimodal exercise to perform exercises of different characteristics, including aerobic exercises, balance exercises and low-load strength exercises for muscle groups, both in the upper quadrant and the lower quadrant. The sessions were structured according to the recommendations of the American College of Sports Medicine (ACSM) 18, with an initial warm-up (2-3 minutes), a main part (8-12 minutes) and a final cool-down and relaxation (5 minutes).
  Interventions: Other: Oncological functional reeducation program

INTERVENTIONS:
Other: Oncological functional reeducation program — It will consist of the following actions:
  1. Prescription of multimodal physical exercise.
  2. Retraining in activities of daily living.

SUMMARY:
In recent years the survival of cancer patients has increased exponentially. But together with that survival, and due to the different oncological treatments, side effects have also increased significantly. Some of these may be tumor asthenia or dyspnea. The latter can represent a serious health problem, with important limitations for individuals. To control this, we consider that the measures used in conventional clinical practice can be implemented, mainly developed through physical exercise. But we believe that not only this is enough, but we also propose an intervention with a comprehensive perspective from the rehabilitative approach, with the aim of integrating education and training of the oncological patient with dyspnea. We propose to combine the intervention with physical exercise with a re-education in the performance of activities of daily living, within a "Functional Oncological Re-education Program", to see if in this way better results are achieved in clinical practice.

That is why we propose to verify the effects produced by the implementation of a multimodal physical exercise program with a specific autonomy recovery program in comparison with an isolated intervention through physical exercise on the functionality and physical performance in cancer patients with dyspnea . To do this, we proposed an experimental, prospective, randomized study using a parallel scheme of fixed assignment with an experimental group and a control group in patients from the Oncology Hospitalization Unit of the Salamanca University Hospital Complex. 44 participants with dyspnea, who were admitted at the time of inclusion, will be selected through a consecutive sampling. After the baseline evaluation, the participants will be randomized into two groups. The subjects of the experimental group will carry out a Rehabilitation Program in addition to the physical exercise carried out in all the participants. The main variable will be the performance of basic activities of daily living (Barthel scale) and the degree of dyspnea (mMRC scale). In addition, physical performance (SPPB), blood oxygen saturation (pulse oximetry), fear / avoidance of movement / TAMPA scale) and quality of life in cancer patients (ECOG) will be assessed. The results of this study could be transferred to the clinic, incorporating them into care protocols for cancer patients with dyspnea.

ELIGIBILITY:
* Inclusion criteria: pathological diagnosis of oncological disease, being admitted at the time of recruitment in the Oncology Unit of CAUSA, presenting dyspnea parameters equal to or greater than "2" points on the Medical Research Council (MRC) scale, a scoring less than 85 points on the Barthel index and having signed an informed consent that indicates the voluntary agreement to participate in the study.
* Exclusion criteria: not having an adequate cognitive state to understand and carry out the orders that are provided (scores lower than 23 points in Mini Mental State Examination, MMSE), present hemoglobin levels lower than 10g / dl, be an active smoker at the time of recruitment.
* Withdrawal criteria: progression of the disease that leads the patient to a terminal situation or death and failure to carry out the follow-up and final evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Dependency level | From the moment of admission to the hospital, until the moment of discharge, an average of 15 days.
  Barthel Index: Measure of physical disability with proven validity and reliability, easy to apply and interpret. Useful to assess functional disability in basic activities of daily living (ABVD). It establishes scores from 0 to 100 in which it quantifies the degree of dependence of the individual.
Level of dyspnea | From the moment of admission to the hospital, until the moment of discharge, an average of 15 days.
  Medical Research Council de Disnea (mMRC): Its objective is to allow the patient to quantitatively grade their own dyspnea visually and easily. Establishes 5 degrees of dyspnea involvement in activities.

SECONDARY OUTCOMES:
Physical performance | From the moment of admission to the hospital, until the moment of discharge, an average of 15 days.
  Short Physical Performance Score (SPPB): The short physical performance battery, validated in our setting for primary health care, is a test specifically designed to predict disabilities and has demonstrated the ability to predict adverse events, dependency, institutionalization, and mortality.
kinesiophobia | From the moment of admission to the hospital, until the moment of discharge, an average of 15 days.
  Tampa Scale for Fatigue Associated Kinesiophobia (TSK-F): scale developed to assess fear of movement related to fatigue / pain, having been validated in cancer patients and chronic fatigue syndrome. The 11-item model (TSK-F-11) will be applied.
Performance status | From the moment of admission to the hospital, until the moment of discharge, an average of 15 days.
  ECOG scale: it is a practical way to measure the quality of life of an oncology patient, whose life expectancy changes over the course of months, weeks and even days. It was designed by the Eastern Cooperative Oncology Group (ECOG) in the United States and validated by the World Health Organization (WHO). The main function of this scale is to objectify the quality of life of the patient or "performance status".
Blood oxygen saturation | From the moment of admission to the hospital, until the moment of discharge, an average of 15 days.
  Pulse oximetry: non-invasive technique that measures the oxygen saturation (Sat O2) of hemoglobin in circulating blood, usually arterial blood, carried out using a pulse oximeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Rodriguez EJ, Gonzalez-Sanchez J, Puente-Gonzalez AS, Recio-Rodriguez JI, Sanchez-Gomez C, Mendez-Sanchez R, Cruz-Hernandez JJ, Rihuete-Galve MI. Specific autonomy recovery programme in a comprehensive rehabilitation on functionality and respiratory parameters in oncological patients with dyspnoea. Study protocol. BMC Nurs. 2021 Jul 5;20(1):120. doi: 10.1186/s12912-021-00633-z. PMID 34225735